CLINICAL TRIAL: NCT04224597
Title: Evaluation of the Presence of Enthesitis in Patients With Acne Vulgaris
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Erol Olcok Corum Training and Research Hospital (Other)
Responsible Party: Principal Investigator, Dilek Eker Büyükşireci, Specialist doctor, Erol Olcok Corum Training and Research Hospital
Other Study IDs: Hitit University
Record Dates: First submitted 2020-01-08; First posted 2020-01-13 (Actual); Last update posted 2020-01-27 (Actual); Status verified 2020-01

CONDITIONS: Enthesitis; Acne Vulgaris; Ultrasonography
Keywords: enthesitis; acne vulgaris; Guess
MeSH Terms: conditions — Acne Vulgaris | interventions — Ultrasonography

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Patients with acne vulgaris: patients with acne vulgaris aged between 18-25 year
  Interventions: Diagnostic Test: ultrasonography
- Healthy controls: healthy controls aged between 18-25 year
  Interventions: Diagnostic Test: ultrasonography

INTERVENTIONS:
Diagnostic Test: ultrasonography — all participants will be determined by ultrasonography.

SUMMARY:
Acne vulgaris is an inflammatory disease of the pilosebaceous unit, affecting about 85% of the young population. In the studies p. acne is a potent stimulator of the release of IFN-gamma (IFN-)) and IL-17 from CD4 + T cells, and the presence of IL-17 + cells in the perifollicular infiltrate has been shown in biopsies of inflammatory acne lesions. Therefore, acne is thought to be a Th17-related disease (1).

This study was aimed to evaluate the presence of enthesitis in patients with acne vulgaris.

DETAILED DESCRIPTION:
Patients with acne vulgaris and healthy controls aged between 18-25 who admitted to Hitit University Erol Olcok Education and Research Hostpital Dermatology policlinic will be icluded. Patients with rheumatic, neurological diseases, history of trauma and previous fractures will be excluded from the study. After all the participants were evaluated by the dermatologist and demographic data will be recorded, the participants will be examined by the physical medicine and rehabilitation specialist and the short form-36 (sf-36), hospital anxiety and depression scale will be completed. Bilateral lower extremity tendon thicknesses and the presence of erosion, bursitis, etc. will be evaluated according to the criteria of Guess (Glasgow Ultrasound Enthesitis Scoring System) and Guess score will be determined for all participants. A total of 48 participants, 24 patients with acne vulgaris and 24 healthy controls, will be included in the study (2).

ELIGIBILITY:
Inclusion Criteira:

* Patients with acne vulgaris and healthy controls aged between 18-25

Exclusion Criteria:

* Participants with rheumatic and neurologic disease, history of trauma ,

Ages: 18 Years to 25 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes
Study Population: Patients with acne vulgaris and healthy controls aged between 18-25
Sampling Method: Probability Sample
Enrollment: 48 (Estimated)
Dates: Start 2020-02-01 (Estimated); Primary Completion 2020-04-01 (Estimated); Study Completion 2020-04-01 (Estimated)

PRIMARY OUTCOMES:
patellar tendon thicknesses of patients with acne vulgaris and healthy controls | 3 months
Ashilles tendon thicknesses of patients with acne vulgaris and healthy controls | 3 months

CONTACTS AND LOCATIONS:
Locations (1):
- Dilek Eker Büyükşireci, Çorum, Central Anatolia, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No